CLINICAL TRIAL: NCT02733432
Title: A Phase 2, Multicenter, Randomized, Active-controlled Study of the Safety and Tolerability of Two Formulations of CD101 Compared to Fluconazole for the Treatment of Moderate to Severe Episodes of Acute Vulvovaginal Candidiasis
Brief Title: RADIANT: CD101 vs Standard of Care in Subjects With Acute Vaginal Yeast Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD101.TP.2.01
Record Dates: First submitted 2016-03-28; First posted 2016-04-11 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2018-03

CONDITIONS: Candidiasis, Vulvovaginal; Mycoses; Yeast Infection; Moniliasis, Vulvovaginal; Vaginitis, Monilial
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Mycoses | interventions — Fluconazole

STUDY DESIGN:
Masking Description: Sponsor blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): CD101 Vaginal Gel (3%) topically self-administered intravaginally as a single dose on days 1 and 2 and for symptomatic relief CD101 External Gel (1%)topically self-applied to external vulva up to twice per day over 72 hours.
  Interventions: Drug: CD101 Vaginal Gel (3%); Drug: CD101 External gel (1%)
- Cohort 2 (Experimental): CD101 Vaginal Ointment (6%) topically self-administered intravaginally as a single dose on day 1 and for symptomatic relief CD101 External Ointment (1%) topically self-applied to external vulva up to twice per day over 72 hours.
  Interventions: Drug: CD101 Vaginal Ointment (6%); Drug: CD101 External ointment (1%)
- Cohort 3 (Active Comparator): Oral fluconazole (150mg) administered on day 1.
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: CD101 Vaginal Gel (3%) — CD101 Vaginal Gel (3%) intravaginally applied topical gel on Days 1 and 2
  Arms: Cohort 1
Drug: CD101 External gel (1%) — CD101 external gel (1%) applied topically twice daily over 72 hours as needed
  Arms: Cohort 1
Drug: CD101 Vaginal Ointment (6%) — CD101 vaginal ointment (6%) intravaginally applied topical ointment on Day 1
  Arms: Cohort 2
Drug: CD101 External ointment (1%) — CD101 external ointment (1%) applied topically twice daily over 72 hours as needed
  Arms: Cohort 2
Drug: Fluconazole — oral fluconazole (150mg) on Day 1
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to determine if two topical formulations of CD101 are safe and effective in the treatment of acute moderate to severe vulvovaginal candidiasis (VVC) compared to oral fluconazole.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, open-label, sponsor-blind, active-controlled, dose-ranging trial of female subjects with an acute moderate to severe episode of vulvovaginal candidiasis. Subjects will be randomized to 1 of 3 treatment arms; CD101 gel, CD101 ointment, or oral fluconazole. After randomization, subjects will be seen on Day 7 (+/-2 days), Day 14 (+/- 2 days), & Day 28 (+/-7 days) to assess therapeutic cure and safety.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe acute vulvovaginal candidiasis (severity score >7)
* positive potassium hydroxide wet preparation for pseudohyphae or budding yeast or positive Becton Dickinson Affirm test or positive vaginal culture for Candida species
* vaginal pH <4.5 for subjects with positive potassium hydroxide wet preparation
* able to give written informed consent

Exclusion Criteria:

* receipt of intravaginal or systemic antifungal therapy within 7 days of randomization
* known or suspected infectious causes of vulvovaginitis other than candidiasis
* history of genital herpes
* planned treatment or surgery during the study period for cervical intraepithelial neoplasia or cervical carcinoma
* need for non-protocol systemic or vaginal antifungal therapy
* history of hypersensitivity or allergic reaction to echinocandins, azoles, or their excipients
* pregnant females
* females who are breast feeding
* women intending to become pregnant during the study period
* recent use of an investigational medicinal product within 28 days or presence of an investigational device at the time of screening
* subjects who use or anticipate use of intravaginal products
* have any condition that the Investigator believes would put the subject at risk for participation or would confound the results of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Incidence of Treatment Emergent Adverse Events [Safety and Tolerability] | Day 28 - 35
  adverse events, clinical chemistry and hematology, pelvic exams

SECONDARY OUTCOMES:
Change in Vulvovaginal Scoring System | Day 7 (+/- 2days)
  Change in clinical signs and subject symptoms of VVC
Change in Vulvovaginal Scoring System | Day 14 (+/- 2days)
  Change in clinical signs and subject symptoms of VVC
Change in Vulvovaginal Scoring System | Day 28 - 35
  Change in clinical signs and subject symptoms of VVC
Mycological Culture | Day 7 (+/- 2days)
  Culture negative for Candida
Mycological Culture | Day 14 (+/- 2days)
  Culture negative Candida
Mycological Culture | Day 28 -35
  Culture negative Candida

CONTACTS AND LOCATIONS:
Overall Officials: Alena Jandourek, MD, Study Director — Cidara Therapeutics
Locations (24):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Precision Trials AZ LLC, Phoenix, Arizona
  - The Women's Clinical, P.A., Little Rock, Arkansas
  - Women's Health Care Research Corp, San Diego, California
  - Olympian Clinical Research, Clearwater, Florida
  - Women's Medical Research, Clearwater, Florida
  - Altus Research Inc, Lake Worth, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Augusta University, Augusta, Georgia
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Tolan Park Clinic, Detroit, Michigan
  - Saginaw Valley Medical Research Group LLC, Saginaw, Michigan
  - Lawrence OB GYN Clinical Research LLC, Lawrenceville, New Jersey
  - Alliance Women's Research Group LLC, Riverside Park, New Jersey
  - ProHEALTH Care Associates, LLP, Port Jefferson, New York
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Hawthorne Medical Research Inc, Winston-Salem, North Carolina
  - Unified Women's Clinical Research - Hickory, Winston-Salem, North Carolina
  - Aventiv Research Inc, Columbus, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - TMC Life Research Inc., Houston, Texas
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Tidewater Clinical Research, Inc, Norfolk, Virginia
  - Seattle Women's Health, Research, Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided